CLINICAL TRIAL: NCT00304954
Title: Treatment of Choroidal Subretinal Neovascularization With Agents Directed Against the Immune Response
Brief Title: Infliximab, Sirolimus and Daclizumab to Treat Age-Related Macular Degeneration
Acronym: AMDB1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 060111; 06-EI-0111 (Other: NEI)
Record Dates: First submitted 2006-03-17; First posted 2006-03-20 (Estimated); Results first posted 2011-04-12 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-11

CONDITIONS: Age-Related Macular Degeneration; Choroidal Neovascularization
Keywords: Age-Related Macular Degeneration; Rapamycin; Remicade; Daclizumab; Immunosuppression; Infliximab; Choroidal Neovascularization; Sirolimus; AMD; Ocular Inflammation
MeSH Terms: conditions — Macular Degeneration; Choroidal Neovascularization | interventions — Daclizumab; Infliximab; Observation; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Intravenous Daclizumab (Active Comparator): Participants randomly assigned to intravenous (IV) daclizumab received 8 mg/kg of IV daclizumab at baseline, then 4 mg/kg of IV daclizumab at Week 2 and then 2 mg/kg of IV daclizumab monthly for the rest of the 6-month study.
  Interventions: Drug: Intravenous Daclizumab
- Intravenous Infliximab (Active Comparator): Participants randomized to IV infliximab received 3 mg/kg of IV infliximab monthly for 6 months.
  Interventions: Drug: Intravenous Infliximab
- Oral Rapamycin (Active Comparator): Participants randomly assigned to rapamycin received 2 mg in capsule form every other day for 6 months.
  Interventions: Drug: Oral Rapamycin
- Observation (Other): Participants randomly assigned to the observation group were given injections of either bevacizumab (1.25 mg/0.05 mL or 2.5 mg/0.1 mL) or ranibizumab (0.5 mg) if they presented with recurrence of intraretinal or subretinal fluid as seen on Stratus Optical Coherence Tomography.
  Interventions: Other: Observation

INTERVENTIONS:
Drug: Intravenous Daclizumab — Participants randomly assigned to intravenous (IV) daclizumab received 8 mg/kg of IV daclizumab at baseline, then 4 mg/kg of IV daclizumab at Week 2 and then 2 mg/kg of IV daclizumab monthly for the rest of the 6-month study.
  Other Names: Zenapax
  Arms: Intravenous Daclizumab
Drug: Intravenous Infliximab — Participants randomized to IV infliximab received 3 mg/kg of IV infliximab monthly for 6 months.
  Other Names: Remicade
  Arms: Intravenous Infliximab
Other: Observation — Participants randomly assigned to the observation group were given injections of either bevacizumab (1.25 mg/0.05 mL or 2.5 mg/0.1 mL) or ranibizumab (0.5 mg) if they presented with recurrence of intraretinal or subretinal fluid as seen on Stratus Optical Coherence Tomography.
  Arms: Observation
Drug: Oral Rapamycin — Participants randomly assigned to rapamycin received 2 mg in capsule form every other day for 6 months.
  Other Names: Sirolimus
  Arms: Oral Rapamycin

SUMMARY:
This study examined whether the anti-inflammatory medicines infliximab, sirolimus or daclizumab, when given with a participant's current therapies, would prevent the growth of new blood vessels in the eye in participants with age-related macular degeneration (AMD).

Participants 55 years of age and older with AMD and drusen larger than 63um may be eligible for this study. Vision in the study eye was between 20/20 and 20/400.

Participants were randomly assigned to one of three treatments - infliximab, sirolimus, or daclizumab - or to observation only. In addition, participants may have been treated by their ophthalmologist as needed for their AMD.

Infliximab and daclizumab were given intravenously (through a vein); infusions were given at enrollment in the study, then at 2 weeks, and then monthly.

Sirolimus was a pill that was taken every other day for the duration of the study. At 6 months, participants were evaluated to see whether continuing treatment would be beneficial.

In addition to treatment or observation, participants underwent the following procedures:

Physical examination at enrollment and 6 months.

Photographs of the back of the eye, fluorescein angiography, indocyanine green angiography and measurement of retinal thickness at enrollment and months 1, 3 and 6.

* Fluorescein angiography evaluated the eye's blood vessels. A yellow dye was injected into an arm vein and traveled to the blood vessels in the eyes. Pictures of the retina were taken using a camera that flashed a blue light into the eye. The pictures show if any dye has leaked from the vessels into the retina, indicating possible blood vessel abnormality.
* Indocyanine green angiography identified feeder vessels that may have supplied abnormal blood vessels. This procedure is similar to fluorescein angiography, but uses a green dye and flashes an invisible light.
* Optical coherence tomography measures retinal thickness. This test shines a light into the eye and produces cross-sectional pictures of the retina. These measurements are repeated during the study to determine whether retinal thickening is getting better or worse, or staying the same.

Tuberculin skin test and chest x-ray at enrollment and 6 months.

Blood tests at enrollment and months 1, 3 and 6.

DETAILED DESCRIPTION:
There has been much interest in the possible role of the immune system in AMD. Experimental models and patient material have, to date, suggested a role for macrophages and complement. This study hypothesized that the underlying mechanism that leads to choroidal neovascularization (CNV) is similar to those at play in atherosclerosis. If this is the case, the investigators believed that CNV treatment should be amenable to new immunomodulatory agents directed against specific parts of the immune system.

After therapy with anti-angiogenic agents not leading to a persistent remission of CNV due to AMD, participants were treated with one of three immunomodulatory agents or were observed in conjunction with their continued anti-angiogenic therapy. Thus the participant continued with the anti-angiogenic therapy they received after randomization. The investigators hypothesized that this combination therapy would inhibit progression of CNV associated with AMD.

This was an open-label, phase II, randomized, single center clinical trial of 18 study participants randomized to receive one of three immunomodulatory agents or was observed in conjunction with their anti-angiogenic therapy.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Understand and sign the institutional review board (IRB)-approved informed consent document for the study.
2. Age greater than 55 years.
3. In the study eye, diagnosis of AMD defined by the presence of drusen larger than 63 microns.
4. Any anti-angiogenic therapy in the study eye within 7 days of beginning immunosuppressive therapy.
5. In the study eye, the participant's study eye vision is between 20/20 and 20/400.
6. In the study eye, the presence of CNV under the fovea determined by the investigators and defined as any one of the following fluorescein angiographic (FA) features:

   1. Early stippled hyperfluorescence of flat retinal pigment epithelium (RPE)and little or mild leakage in the late frames of the fluorescein (occult).
   2. Irregular elevation of the RPE that does not exhibit discrete or bright hyperfluorescence in the early transit phase of the angiogram. Stippled hyperfluorescence may be present. Late frames may show persistent fluorescein staining or leakage within a sensory retinal detachment overlying this area (occult).
   3. Late-phase leakage of undetermined source with leakage at the level of the RPE in the late-phase frames of the angiogram in which the source of the late leakage cannot be determined from earlier-phase frames of the angiogram (occult).
   4. A well-demarcated area of bright hyperfluorescence in the early phase of the angiogram with leakage through the mid- and late-phase frames which obscures the boundaries of the area (classic).
7. For all CNV lesions considered to have occult CNV with no classic CNV, one of the following criteria must be met:

   1. A documented loss of visual acuity (5 or more letters of best-corrected visual acuity if both measurements are made using an Early Treatment for Diabetic Retinopathy Study (ETDRS) chart or, a doubling of the visual angle if Snellen acuities are available from either an outside referral center or within the participating center (e.g., 20/80 to 20/160) a doubling of the visual angle is required because of the measurement variability of Snellen acuities).

      OR
   2. Documented FA evidence of a 10% increase in the lesion greatest linear dimension over the 3 months prior to enrollment.

      OR
   3. Documented blood associated with CNV.
8. The greatest linear dimension of the entire lesion (classic CNV, occult CNV and any features that could obscure the identification of classic or occult CNV) has to be less than or equal to 5400 microns in greatest linear dimension on the retina as measured by the treating ophthalmologist.
9. Retinal photographs and angiography of sufficient quality, allowing assessment of the macular area according to standard clinical practice, can be obtained.
10. Women of childbearing potential must not be pregnant or lactating, must have a negative pregnancy test at screening and must be practicing an adequate method of birth control. Acceptable methods of birth control include intrauterine device (IUD); oral, dermal, implanted or injected contraceptives; tubal ligation; and barrier methods with spermicide.
11. Willingness to comply with the protocol.

EXCLUSION CRITERIA:

1. CNV, in the study eye, associated with other ocular diseases such as pathologic myopia, ocular histoplasmosis or posterior uveitis, etc.
2. Presence of geographic atrophy under the fovea in the study eye.
3. Evidence of retinal angiomatous proliferation as suspected by the presence of intraretinal hemorrhage, intraretinal leakage, adjoining serous pigment epithelial detachment (PED) or the presence of a connecting retinal vessel.
4. The presence of a chorio-retinal anastomosis.
5. Decreased vision, in the study eye, due to retinal disease not attributable to CNV, such as nonexudative forms of AMD, geographic atrophy, inherited retinal dystrophy, uveitis or epiretinal membrane. Participants who have any additional ocular diseases that have irreversibly compromised or, during follow-up, could likely compromise the visual acuity (VA) of the study eye including amblyopia, anterior ischemic optic neuropathy, clinically significant diabetic macular edema, severe non-proliferative diabetic retinopathy, or proliferative diabetic retinopathy.
6. Decreased vision, in the study eye, due to significant media opacity such as corneal disease or cataract, or opacity precluding photography of the retina; a tear (rip) of the RPE; a vitelliform-like lesion of the outer retina (e.g., as in pattern dystrophies or basal laminar drusen), idiopathic parafoveal telangiectasis, or central serous retinopathy.
7. Presence of fibrosis, hemorrhage, pigment epithelial detachments and other hypofluorescent lesions obscuring greater than 50% of the CNV lesion.
8. History of other systemic antiangiogenic treatment or treatment for CNV (not including photodynamic therapy and pegaptanib sodium injections) in the study eye with transpupillary thermotherapy or other local treatment (such as submacular surgery). Previous laser photocoagulation therapy is acceptable, provided it was not subfoveal.
9. Participant with a known underlying systemic disease with evidence of serious or potentially lethal uncontrolled active disease in one or more extraocular organ systems for which a defined effective medical regimen is indicated.
10. Participant with a corneal melting, necrotizing keratitis, or impending vision loss.
11. Participants with history of allergy to/or exposure to mouse protein.
12. Participant with scleritis of infectious etiology.
13. Participant receiving any other investigational therapy or another anti-tumor necrosis factor (TNF) agent that would interfere with the ability to evaluate the safety or efficacy of infliximab.
14. Participant has significant active infection requiring hospitalization.
15. Participant with multiple sclerosis.
16. Participant has severe (class 3/4) congestive heart failure.
17. Participant has a history of cancer within the past 5 years other than basal or squamous cell carcinoma.
18. Participant is pregnant or lactating.
19. Participant with posterior scleritis.
20. Participant has evidence of liver disease (any etiology). History of moderate to severe abnormal liver function, unless documented evidence of normal liver enzymes is provided.
21. Participant has positive PPD (tuberculosis test) unless cleared by Internal Medicine.
22. Participant has positive Chest X-ray showing acute pulmonary disease.
23. Participant has unexplained hematuria.
24. Participant has a history of alkylating therapy use.
25. Current exam evidence of ocular toxoplasmosis; pseudoexfoliation; external ocular infection, including conjunctivitis; chalazion; significant blepharitis; or aphakia in the study eye (pseudophakic participants are eligible).
26. Intraocular surgery (including lens replacement surgery) within 6 weeks prior to randomization.
27. Recent history of (within the last 6 months), or current acute ocular or periocular infection (including any history of ocular herpes zoster or simplex).
28. Known hypersensitivity/allergy to verteporfin, porfimer sodium, or other porphyrins, porphyria or other porphyrin sensitivity, or hypersensitivity to sunlight or bright artificial light. Participation in any other clinical study or are receiving, or have received any experimental systemic treatment for AMD (e.g., retinoic acid, thalidomide). Local therapy for AMD is permitted.
29. Medical problems that make consistent follow-up over the treatment period unlikely (e.g., stroke, severe myocardial infarction (MI), end stage malignancy), any contraindications to performing the necessary diagnostic studies (i.e., known allergy to fluorescein dyes etc.), or in general a poor medical risk because of other systemic diseases or active uncontrolled infections.
30. Participant has a history of moderate to severe abnormal liver function, unless documented evidence of normal liver enzymes is provided.
31. Participant has a history of active pulmonary tuberculosis.
32. Participant has a history of active viral hepatitis.
33. Participant has chronic continued Ketoconazole use.

Ages: 55 Years to 92 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2006-02; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Nussenblatt, MD, MPH, Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Aeberli D, Oertle S, Mauron H, Reichenbach S, Jordi B, Villiger PM. Inhibition of the TNF-pathway: use of infliximab and etanercept as remission-inducing agents in cases of therapy-resistant chronic inflammatory disorders. Swiss Med Wkly. 2002 Jul 27;132(29-30):414-22. doi: 10.4414/smw.2002.10031. PMID 12428187
- [Background] Antoni C, Dechant C, Hanns-Martin Lorenz PD, Wendler J, Ogilvie A, Lueftl M, Kalden-Nemeth D, Kalden JR, Manger B. Open-label study of infliximab treatment for psoriatic arthritis: clinical and magnetic resonance imaging measurements of reduction of inflammation. Arthritis Rheum. 2002 Oct 15;47(5):506-12. doi: 10.1002/art.10671. PMID 12382299
- [Background] Bian ZM, Elner SG, Strieter RM, Kunkel SL, Lukacs NW, Elner VM. IL-4 potentiates IL-1beta- and TNF-alpha-stimulated IL-8 and MCP-1 protein production in human retinal pigment epithelial cells. Curr Eye Res. 1999 May;18(5):349-57. doi: 10.1076/ceyr.18.5.349.5353. PMID 10372996
- [Result] Nussenblatt RB, Byrnes G, Sen HN, Yeh S, Faia L, Meyerle C, Wroblewski K, Li Z, Liu B, Chew E, Sherry PR, Friedman P, Gill F, Ferris F 3rd. A randomized pilot study of systemic immunosuppression in the treatment of age-related macular degeneration with choroidal neovascularization. Retina. 2010 Nov-Dec;30(10):1579-87. doi: 10.1097/IAE.0b013e3181e7978e. PMID 20847709

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at the Clinical Center, NIH. A total of 13 participants met the eligibility criteria for the study and were enrolled from September 2006 to May 2008.
Period: Overall Study
Arm/Group | Intravenous Daclizumab | Intravenous Infliximab | Oral Rapamycin | Observation
Started | 4 | 3 | 3 | 3
Completed | 3 | 3 | 2 | 3
Not Completed | 1 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intravenous Daclizumab | Intravenous Infliximab | Oral Rapamycin | Observation | Total
Number analyzed (Participants) | 4 | 3 | 3 | 3 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 0 | 0 | 1
  >=65 years | 3 | 3 | 3 | 3 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 79 (13) | 77 (8) | 78 (7) | 87 (4) | 80 (9)
Gender [Count of Participants; unit: Participants]
  Female | 4 | 2 | 3 | 3 | 12
  Male | 0 | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 3 | 3 | 13

OUTCOME MEASURES:

1. Primary Outcome: Monthly Rates of Anti-VEGF (Vascular Endothelial Growth Factor) Injections
Time Frame: 24 Weeks
Measure: Median (Full Range); unit: Injections per Month
Arm/Group | Intravenous Daclizumab | Intravenous Infliximab | Oral Rapamycin | Observation
Number analyzed (Participants) | 4 | 3 | 3 | 3
Injections per Month | 0.42 [0.34 to 0.83] | 0.83 [0.5 to 1] | 0.34 [0.29 to 0.5] | 0.83 [0.5 to 1]

2. Secondary Outcome: Changes in Best-corrected Visual Acuity (BCVA) as Measured by the Standard Early Treatment Diabetic Retinopathy Study (ETDRS) Protocol From Baseline to 24 Weeks
Description: The values in the table represent the denominator for the visual acuity in feet. A value of 20 represents "normal" 20/20 vision while increasing values for the denominator represent worsening vision.
Time Frame: Baseline and 6 months (24 weeks) - Baseline and 3.5 months for Patient 7
Measure: Number; unit: Feet
Arm/Group | Baseline Vision - Study Eye | Sixth-Month Vision - Study Eye | Baseline Vision - Fellow Eye | Sixth-Month Vision - Fellow Eye
Number analyzed (Participants) | 13 | 13 | 13 | 13
Feet
  Rapamycin Patient 1 | 40 | 25 | 400 | 640
  Rapamycin Patient 7 (Baseline and 3.5 months) | 63 | 50 | 640 | 640
  Rapamycin Patient 12t | 32 | 32 | 32 | 32
  Daclizumab Patient 3 | 40 | 40 | 40 | 32
  Daclizumab Patient 8 | 32 | 32 | 32 | 32
  Daclizumab Patient 9 | 250 | 250 | 63 | 40
  Daclizumab Patient 13 | 50 | 40 | 25 | 20
  Infliximab Patient 2 | 40 | 32 | 63 | 125
  Infliximab Patient 6 | 250 | 800 | 63 | 80
  Infliximab Patient 10 | 50 | 32 | 125 | 125
  Observation Patient 4 | 63 | 63 | 40 | 25
  Observation Patient 5 | 50 | 25 | NA — Vision too low to arrive at value. Counting fingers used instead. | NA — Vision too low to arrive at value. Counting fingers used instead.
  Observation Patient 11 | 32 | 50 | 200 | 63

3. Secondary Outcome: Changes in Retinal Thickness as Measured by Optical Coherence Tomography (OCT) From Baseline to 24 Weeks
Time Frame: Baseline and 6 months (24 weeks) - Baseline and 3.5 months for Patient 7
Measure: Number; unit: Microns
Arm/Group | Baseline OCT - Study Eye | Sixth-Month OCT - Study Eye | Baseline OCT - Fellow Eye | Sixth-Month OCT - Fellow Eye
Number analyzed (Participants) | 13 | 13 | 13 | 13
Microns
  Rapamycin Patient 1 | 234 | 230 | 211 | 203
  Rapamycin Patient 7 (Baseline and 3.5 months) | 361 | 239 | 242 | 186
  Rapamycin Patient 12t | 327 | 264 | 226 | 205
  Daclizumab Patient 3 | 216 | 189 | 352 | 206
  Daclizumab Patient 8 | 185 | 208 | 218 | 149
  Daclizumab Patient 9 | 297 | 196 | 215 | 210
  Daclizumab Patient 13 | 329 | 344 | 305 | 317
  Infliximab Patient 2 | 205 | 177 | 190 | 181
  Infliximab Patient 6 | 290 | 243 | 262 | 252
  Infliximab Patient 10 | 291 | 288 | 453 | 347
  Observation Patient 4 | 229 | 196 | 189 | 171
  Observation Patient 5 | 426 | 225 | 270 | 213
  Observation Patient 11 | 318 | 305 | 158 | 169

ADVERSE EVENTS:
Time Frame: February 14, 2006 through December 30, 2009
Arm/Group | Intravenous Daclizumab | Intravenous Infliximab | Oral Rapamycin | Observation
Serious Adverse Events (participants affected / at risk) | 1/4 | 0/3 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3 | 3/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intravenous Daclizumab (N=4) | Intravenous Infliximab (N=3) | Oral Rapamycin (N=3) | Observation (N=3)
Episode of right sided numbness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intravenous Daclizumab (N=4) | Intravenous Infliximab (N=3) | Oral Rapamycin (N=3) | Observation (N=3)
Decreased Albumin (Blood and lymphatic system disorders) | 4 (5) | 2 (2) | 1 (1) | 1 (1)
Elevated Blood Urea Nitrogen (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Elevated C02 (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Decreased Total Protein (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Pruritus on Torso and Upper Arms (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased Phosphorus (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Elevated Phosphorus (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Elevated Chloride (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Elevated Red Blood Cell Count (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Fecal Incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stress Incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Blurred Vision (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ankle Edema (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Elevated Ethrocyte Sedimentation Rate (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lacrimal Gland Lesion (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tingling Hands (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthritis Hands (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Leg Cramps (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Elevated Low-density Lipoprotein (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Elevated Cholesterol (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Decreased Hematocrit (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Elevated Basophils (Blood and lymphatic system disorders) | 3 (3) | 2 (2) | 0 (0) | 2 (2)
Elevated Bilirubin (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Migraine Symptoms (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Elevated Eosinophils (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Aortic Anneurysm (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Elevated White Blood Cells in Urine (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Decreased Red Cell Distribution Width (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Elevated Uric Acid (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Elevated Lymphocytes (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Pigmented Papule on Eyelid (Eye disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Seborrheic Keratoses Eyelid (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased Sodium (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Elevated White Blood Cell Count (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Elevated Neutrophils (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Iris Nevi (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vitreous Syneresis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Elevated Red Blood Cells in Urine (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Ptosis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Elevated Potassium (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vitreous Detachment (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Elevated Alanine Transaminase (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Elevated Aspartate Aminotransferase (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Elevated Hematocrit (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Elevated Hemoglobin (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Elevated Thyroid Stimulating Hormone (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fluttering in Chest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Leukocyte Esterase in Urine (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Scratchy Throat (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Vision Decrease (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Elevated Monocytes (Blood and lymphatic system disorders) | 3 (3) | 1 (1) | 2 (2) | 0 (0)
Flu (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypercholesteremia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Irregular Heart Rate (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Electrolyte Imbalance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metamorphosia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weakness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Foot Ulcer (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Achiness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper Respiratory Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Elevated Magnesium (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Elevated Lactate Dehydrogenase (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased Chloride (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased Hemoglobin (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Decreased Magnesium (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased Low-density Lipoprotein (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased Red Blood Cell Count (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Elevated Glucose (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased Neutrophils (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laryngitis (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Discomfort Defacating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Runny Nose (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased Uric Acid (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Elevated Lipids (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Shoulder Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Polymialgia Rheumatica (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased Creatinine Kinase (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased Eosinophils (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased Alkaline Phosphatase (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased Neutrophils (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No